CLINICAL TRIAL: NCT02216305
Title: Prospective and Randomized Trial Comparing Doppler-Guided Transanal Hemorrhoid Artery Ligation With Recto-anal Repair (HAL-RAR) Versus Excisional Hemorrhoidectomy for the Treatment of Grade III-IV Hemorrhoids
Brief Title: HAL-RAR Versus Hemorrhoidectomy in the Treatment of Grade III-IV Hemorrhoids. Prospective, Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Plató (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAL-RAR Plató 2.0
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Hemorrhoids; Pain, Postoperative
Keywords: HAL-RAR; Hemorrhoids; Hemorrhoid artery ligation; Anal repair; Quality of Life; Postoperative Complications
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative; Postoperative Complications | interventions — Hemorrhoidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemorrhoidectomy (Active Comparator): Open hemorrhoidectomy may include one to three anal cushions and made according to the Milligan-Morgan technique, with resection of the anal cushion and the external hemorrhoidal epidermal component using electrocautery and ligation of the hemorrhoidal base with absorbable suture
  Interventions: Procedure: Hemorrhoidectomy
- HAL-RAR (Active Comparator): Hemorrhoidal artery ligation and rectoanal repair will be performed with the AMI minimally invasive surgery device HAL/RAR, and consist in the ligation of the terminal branches of the superior rectal artery with 2-0 absorbable polyglycolic acid suture after identifying the blood flow approximately 3 cm above the dentate line by using Doppler guidance. Subsequently, a running suture was added from the suture point to 5 mm above the dentate line to lift the prolapsing hemorrhoid. Other procedures will not be associated.
  Interventions: Procedure: HAL-RAR

INTERVENTIONS:
Procedure: Hemorrhoidectomy — Open hemorrhoidectomy may include one to three anal cushions and made according to the Milligan-Morgan technique, with resection of the anal cushion and the external hemorrhoidal epidermal component using electrocautery and ligation of the hemorrhoidal base with absorbable suture
  Arms: Hemorrhoidectomy
Procedure: HAL-RAR — Hemorrhoidal artery ligation and rectoanal repair will be performed with the AMI minimally invasive surgery device HAL/RAR, and consist in the ligation of the terminal branches of the superior rectal artery with 2-0 absorbable polyglycolic acid suture after identifying the blood flow approximately 3 cm above the dentate line by using Doppler guidance. Subsequently, a running suture was added from the suture point to 5 mm above the dentate line to lift the prolapsing hemorrhoid. Other procedures will not be associated.
  Other Names: Hemorrhoid Artery Ligation and Rectoanal Repair
  Arms: HAL-RAR

SUMMARY:
HYPOTHESIS

1. HAL- RAR causes a lower immediate postoperative pain compared with excision hemorrhoidectomy.
2. HAL - RAR achieves similar immediate and long term results compared to the excision hemorrhoidectomy in the control of hemorrhoidal symptoms.
3. The complication rate of HAL- RAR is low and similar to excision hemorrhoidectomy.

OBJECTIVES

1. Compare postoperative pain of both techniques.
2. Assess the short and long-term control of hemorrhoidal symptoms by HAL- RAR technique, and compare the results with those of the excision hemorrhoidectomy.
3. Evaluate and compare the rate of complications of both techniques.
4. Assess the quality of life of patients before and after treatment.

DETAILED DESCRIPTION:
The classic surgical treatment of hemorrhoidal disease is the excisional hemorrhoidectomy, that consist in the surgical removal of one or more hemorrhoidal cushion, it is considered a safe, radical and definitive treatment; however, it is not exempt of complications and the postoperative pain is considerable. During the last two decades the concept of treatment has evolved to control hemorrhoidal symptoms with less invasive techniques, such as hemorrhoidal bands, arterial ligation Doppler guided hemorrhoidal and more recently, the association of anorectal repair or mucopexia for treating hemorrhoidal mucosal prolapse .

MATERIAL AND METHODS

The trial was subjected to evaluation and accepted by the Ethics Committee of the Fundació Unió Catalana d'Hospitals (Catalonian Union of Hospitals Foundation).

All patients with grade III and IV hemorrhoids that are eligible for surgical treatment with both methods who agree to participate in the study, will be included in the prospective randomized trial. All patients will be required to sign the specific informed consent.

Patients who are suitable for treatment with both techniques will be randomly assigned to the surgical technique.

Inclusion criteria:

1. Patients with symptomatic grade III or IV hemorrhoids (bleeding, pain, itching, soiling or prolapse) that are eligible for surgical treatment with both methods.

Exclusion criteria:

1. Associated recto-anal pathology such as acute thrombosed hemorrhoid, anal fissure, perianal fistula, perianal abscess, rectal prolapse, fecal incontinence or anal stenosis.
2. Prior anorectal surgery .
3. Systemic pathology that could alter the outcome of the surgery as coagulopathies, chronic pain with continued consumption of analgesics.
4. Age younger than 18 or older than 80 years, socio-pathology or inability to understand the study objectives.

All surgeries are performed on an outpatient basis under regional anesthesia and sedation for the same team of three surgeons. Preoperative preparation consists of a cleansing enema and no prophylactic antibiotics will be administered.

Both techniques will be performed in "Jack -Knife" position. The open hemorrhoidectomy may include one to three anal cushions and made according to the Milligan-Morgan technique, with resection of the anal cushion and the external hemorrhoidal epidermal component using electrocautery and ligation of the hemorrhoidal base with absorbable suture. Once completed hemorrhoidectomy a perianal block is performed with bupivacaine/epinephrine.

Hemorrhoidal artery ligation and rectoanal repair will be performed with the AMI minimally invasive surgery device HAL/RAR, and consist in the ligation of the terminal branches of the superior rectal artery with 2-0 absorbable polyglycolic acid suture after identifying the blood flow approximately 3 cm above the dentate line by using Doppler guidance. Subsequently, a running suture was added from the suture point to 5 mm above the dentate line to lift the prolapsing hemorroid. Other procedures will not be associated, if necessary, the patient will be excluded from the study .

The patient will be discharged if adequate pain control, oral tolerance and spontaneous diuresis is achieved, and after examination by the surgeon in order to discard immediate complications. The ambulatory treatment consists of an osmotic laxative (magnesium hydroxide ), oral analgesia with paracetamol/tramadol ( 325mg/37.5mg ) every 6 hours and Dexketoprofen (25 mg) every 8 hours, metamizol (575 mg) may be associated every 8 hours if pain. In case of persistent pain, the patient will be examined in emergency room.

EVALUATION OF RESULTS A power analysis was performed to assess the study sample size. Choosing a power of 0.8 and a confidence interval of 95% α-error of 0.05, we calculated that 20 patients were needed in each arm.

All patients will be evaluated with a validated questionnaire of 36 questions on quality of life ( SF-36 ) and specific questions about specific symptoms of hemorrhoidal disease (pain, itching , bleeding, soiling and hemorrhoidal prolapse reduction ). The questionnaire will be answered before the intervention, after six and twelve months of follow up.

All patients will complete a diary testing global postoperative pain every day, measured on a numerical scale from 0 to 10 during the first 15 days.

The patients will be assessed on the day of discharge and at 7, 14, and 30 postoperative days. The patients will be evaluated at 6, 12 and 24 postoperative months in the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic grade III or IV hemorrhoids (bleeding, pain, itching, soiling or prolapse) that are eligible for surgical treatment with both methods.

Exclusion Criteria:

* Associated recto-anal pathology such as acute thrombosed hemorrhoid, anal fissure, perianal fistula, perianal abscess, rectal prolapse, fecal incontinence or anal stenosis.
* Prior anorectal surgery .
* Systemic pathology that could alter the outcome of the surgery as coagulopathies, chronic pain with continued consumption of analgesics.
* Age younger than 18 or older than 80 years, socio-pathology or inability to understand the study objectives

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Immediate postoperative pain | up to first 15 postoperative days
  All patients will complete a diary testing global postoperative pain every day, measured on a numerical scale from 0 to 10 during the first 15 days.

SECONDARY OUTCOMES:
Long-term control of hemorrhoidal symptoms | 1, 6, 12 and 24 months after surgery
  Specific symptoms of hemorrhoidal disease (pain, itching , bleeding, soiling and hemorrhoidal prolapse reduction) will be evaluated. Te patient will mark in a questionaire the options "yes" or "no" for each item.

OTHER OUTCOMES:
SF-36 Quality of life score | Preoperative, 6 and 12 months after surgery
  All patients will be evaluated with a validated questionnaire of 36 questions on quality of life ( SF-36 )

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Carvajal, Dr, Principal Investigator — Hospital Plató Barcelona
Locations (1):
- Hospital Plató, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johanson JF, Sonnenberg A. The prevalence of hemorrhoids and chronic constipation. An epidemiologic study. Gastroenterology. 1990 Feb;98(2):380-6. doi: 10.1016/0016-5085(90)90828-o. PMID 2295392
- [Background] Elmer SE, Nygren JO, Lenander CE. A randomized trial of transanal hemorrhoidal dearterialization with anopexy compared with open hemorrhoidectomy in the treatment of hemorrhoids. Dis Colon Rectum. 2013 Apr;56(4):484-90. doi: 10.1097/DCR.0b013e31827a8567. PMID 23478616